CLINICAL TRIAL: NCT02306551
Title: Well Being And Resilience: Mechanisms of Transmission of Health and Risk in Parents With Complex Mental Health Problems and Their Offspring
Brief Title: Well Being And Resilience: Mechanisms of Transmission of Health and Risk
Acronym: WARM
Status: Completed | Type: Observational
Sponsor: Susanne Harder (Other)
Collaborators: University of Glasgow (Other); Psychiatric Research Unit, Psychiatry, Region Zealand, Denmark (Unknown); Region of Southern Denmark (Other)
Responsible Party: Sponsor-Investigator, Susanne Harder, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: DFF-1319-00103
Record Dates: First submitted 2014-11-12; First posted 2014-12-03 (Estimated); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Psychotic Disorder; Bipolar Disorder; Depressive Disorder
Keywords: Offspring; Attachment; Risk development; Resilience
MeSH Terms: conditions — Psychotic Disorders; Bipolar Disorder; Depressive Disorder | interventions — Biological Products

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Psychotic Disorder: Biological and psycho-social risk and resilience factors
  Interventions: Other: Biological and psycho-social risk and resilience factors
- Bipolar Disorder: Biological and psycho-social risk and resilience factors
  Interventions: Other: Biological and psycho-social risk and resilience factors
- Depressive Disorder: Biological and psycho-social risk and resilience factors
  Interventions: Other: Biological and psycho-social risk and resilience factors
- Non-psychiatric Control: Biological and psycho-social risk and resilience factors
  Interventions: Other: Biological and psycho-social risk and resilience factors

INTERVENTIONS:
Other: Biological and psycho-social risk and resilience factors — Naturalistic study, no active intervention or exposure is administered

SUMMARY:
The purpose of this study is to establish a cohort of pregnant women with severe mental disorder and to identify biological and psycho-social transmission mechanisms involved in the development of 'risk' and 'resilience' in the offspring. It is assumed that both 'resilient' and 'risk' development in offspring are caused by a complex interaction between multiple biological, psychological and social factors. The project focuses specifically on exploring the impact of physiological stress-sensitivity, attachment, care-giving and the familial and social context for care-giving. Previous studies support these factors as important for the development of these infants, but systematic research using a prospective design is needed to strengthen evidence and elucidate the importance of these factors in more detail. The interaction over time of physiological stress-sensitivity, attachment, care-giving and the familial and social context for care-giving are evaluated in terms of the evolution of very early indicators of developmental risk and resilience in infants with a known highly increased risk for developing a mental disorder.The findings of the study may potentially lead to more specific targets for preventive interventions, which can improve developmental outcome for these infants.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with Psychotic Disorder (DSM-5: Delusional Disorder (297.1)
* Schizophreniform Disorder (295.4), Schizophrenia (295.90), Schizoaffective Disorder (295.70)
* Brief Psychotic Disorder (298.8) Other specified schizophrenia spectrum and other psychotic disorder (298.8), Unspecified schizophrenia spectrum and other psychotic disorder (298.9) )
* Lifetime diagnosis of DSM-5 Bipolar I and II Disorder (296.89)
* Diagnosis of DSM-5 Major Depressive Disorder current single episode (current 296.22 - 296.25) or recurrent episode (296.32 - 296.35)
* Non-psychiatric control group defined as mothers without any history of treatment or admission for a psychiatric disorder or drug or alcohol addiction.
* Partners of participating women with an expected care-giving role in relation to the infant will also be eligible for participation in the study.
* Infants of participating pregnant women will be included from birth.

Exclusion Criteria:

* Unable to provide informed consent to participate
* Unable to speak English or Danish because of the requirement to complete assessments,
* Miscarriage.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women referred to maternity services or psychiatric services in Denmark in Region Zealand and Region Southern Denmark, in Scotland from NHS Greater Glasgow and Clyde
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2014-09; Primary Completion 2020-08 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Infant attachment as measured by Strange Situation Procedure (Ainsworth et al. 1978) | At infant 52 weeks of age
  Strange Situation Procedure is a structured observation. The infant is videotaped in a playroom during a series of eight structured 3-min episodes involving the baby, the mother, and a female stranger. During the observation the mother leaves and rejoins the infant twice, first leaving the infant with the female stranger, then leaving the infant alone to be rejoined by the stranger. The procedure is designed to be mildly stressful in order to increase the intensity of activation of the infant's attachment behavior. Videotapes are coded for four attachment classifications: secure, avoidant, ambivalent-resistant/dependent and disorganised.

SECONDARY OUTCOMES:
Infant neurobehavioral outcome as measured by Neonatal Intensive Care Unit Neurobehavioral Scale, NNNS, (Lester & Tronick, 2005) | 1-7 days and 4 weeks
  NNNS is a 30-minute, 128-item assessment of neurologic, behavioural, and stress/abstinence signs that evaluates the full range of infant neurobehavior. It has 12 summary scales: habituation, attention, arousal, regulation, number of handling procedures, quality of movement, excitability, lethargy, number of non-optimal reflexes, number of asymmetric reflexes, hypertonicity, and hypotonicity and an additional stress/abstinence scale.
Infant development as measured by Bayley's scales for infant development 3rd edition (BSID-III-R, Bayley, 2006) | 16 and 52 weeks of infant age
  The BSID III-R is a structured observation test assessing cognition, language and motor skills.
Infant stress exposure and physiological stress-sensitivity as measured by hair and salivary cortisol | 1-7 days (hair only) 4 (Saliva only), 16 and 52 weeks of infant age
  Saliva samples are collected before and 20 and 40 minutes after NNNS (4 weeks), still-face procedure (16 weeks) and Strange Situation Procedure (52 weeks)
Infant social-interactive behavior as measured by Coding Interactive Behavior, CIB (Ruth Feldman, 2012) | 1-7 days, 4 and 16 weeks
  CIB is a global measure that looks at parent-child and dyadic affective states and interactive styles. Independent behavioral codes are aggregated into eight higher order constructs: The three child constructs are engagement involvement, withdrawal, and compliance; and the two dyadic constructs are dyadic reciprocity and dyadic negative states.

OTHER OUTCOMES:
Maternal symptom severity as measured by Positive and Negative Syndrome Scale, PANSS, Kay et al.1989, The Montgomery Asberg Depression Rating Scale, MADRS, Montgomery and Asberg, 1979. The Bech-Rafaelsen Mania Rating Scale, BRMRS, Bech et al. 1979. | at baseline before birth of the child and at 1-7 days, 4, 16 and 52 weeks of infant age.
  PANSS, MADRS and BRMRS are rating scales based on a semistructured interview. PANSS 5-factor model assesses the presence or absence of positive, negative, disorganisation, excitement and emotional distress symptoms (van der Gaag et al., 2006). MADRS assesses the presence and severity of 10 core symptoms of depression. BRMRS assesses the presence and severity of 11 core symptoms of hypomania/mania
Parental social risk status as measured by Adverse Childhood Experiences Study Questionnaires (ACES) (Felitti et al., 1998) (trauma, mothers only), work status and level of education | at baseline before birth of the infant
  ACES is a 25-item self report measure that assesses exposure to childhood emotional, physical, or sexual abuse, and household dysfunction during childhood.
Maternal stress-exposure and stress-sensitivity measured by hair and saliva cortisol | During pregnancy and at infant 16 and 52 weeks of age
Parental attachment assessed by The Adult Attachment Interview (AAI, George, Kaplan & Main, 1987) (mothers only), The Adult Attachment Projective (AAP, George & West, 2012) and Psychosis Attachment Measure (PAM, Berry, Wearden & Barrowclough, 2006) | At baseline before birth of the infant
  AAI is a semi-structured interview, consisting of 20 questions and probes, allowing categorisation of an adult individual's state of mind with regard to attachment. (i.e. Secure, Dismissing and Preoccupied, Unresolved and Cannot Classify) The Adult Attachment Projective (AAP, George & West, 2012) consists of eight drawings of attachment situations dealing with illness, solitude, separation, loss, and abuse, along with one neutral scene, A narrative depiction of these drawings is transcribed and coded for attachment representation i.e.. secure, dismissing, preoccupied, or unresolved. PAM, is a self- report questionnaire assessing two dimensions of attachment, anxious and avoidant.
Parental caregiving representation as assessed by Prenatal Care-giving Experiences Questionnaire (PCEQ, Brennan, George, & Solomon, 2013) Care-giving Experiences Questionnaire (CEQ, Brennan, George & Solomon, 2013) | at baseline (PCEQ), 1-7 days, 4,16 and 52 weeks (CEQ)
  PCEQ, and CEQ assesses defensive processing associated with patterns of care-giving representation (George & Solomon, 2008). i.e. flexible integration, deactivation, cognitive disconnection and dimension of care-giving dysregulation as related to infant's secure, avoidant, ambivalent-resistant/dependent and disorganised attachment respectively.
Maternal caregiving behavior as assessed by AMBIANCE (Lyons-Ruth, Bronfmann, & Parson, (1999). Coding Interactive Behavior, CIB (Ruth Feldman, 2012) | 1-7 days, 4 weeks (CIB), 16 and 52 weeks (AMBIANCE)
  The AMBIANCE measure is used to code disrupted caregiver behaviour during videotaped caregiver-infant interactions. The five dimensions of the AMBIANCE coding are: affective communication errors, role/boundary confusion, fearful/disorientation, intrusive/negative, and withdrawing behaviour. CIB is a global measure that looks at parent-child and dyadic affective states and interactive styles. Independent behavioral codes are aggregated into eight higher order constructs: The three adult constructs are sensitivity, intrusiveness, and limit-setting.
Paternal caregiving behavior as assessed by CIB | 16 weeks
  CIB is a global measure that looks at parent-child and dyadic affective states and interactive styles. Independent behavioral codes are aggregated into eight higher order constructs: The three adult constructs are sensitivity, intrusiveness, and limit-setting.
Paternal symptom severity as assessed by Brief Symptom Severity (BSI-53,Derogatis & Melisaratos, 1983) | At baseline before birth of the infant
  BSI-53 is a 53 item self-report inventory.
Parental diagnosis as assessed by Structured Clinical Interview for DSM-5 (SCID) psychosis module (mothers). Structured Assessment of Personality Abbreviated Scale (SAPAS, Moran et al 2003) | At baseline before birth of the infant
  SAPAS is an eight-item screening interview for personality disorder.
Cognitive functioning as assessed by Reynolds Intellectual Screening Test (RIST, Reynolds, Kamphaus and Raines, 2012) | At baseline before birth of the infant
  RIST is a screening measure of general intelligence
Social functioning and support as assessed by Global Assessment of Functioning, GAF(DSM-IV). Significant Other Scale (SOS, Power, Chanpion & Aris) | At baseline and 4, 16 and 52 weeks
  SOS determines two main areas of social support, emotional support and practical support.
Perceived stress as assessed by The Perceived Stress Scale (PSS) | At baseline and at 16 and 52 weeks
  Questions evaluate experiences of life being unpredictable, uncontrollable and distressing during the previous 30 days, and whether the respondent has been feeling nervous or stressed.
Parenting Stress Index, 3rd Edition Short Form (PSI/SF) | At 16 weeks
  Questions assess level of stress related to the parental role
Parental Alliance Measure | At 16 weeks
  Questions assess the parenting aspects of the marital relationship.
ASQ-SE | 52 weeks
  Ages And Stages Questionnaire Social-Emotional

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Harder, PhD, Principal Investigator — Department of Psychology, University of Copenhagen, Denmark; Andrew Gumley, PhD, Principal Investigator — University of Glasgow
Locations (3):
- Denmark (2):
  - Department of child and adolescent mental health Odense, Research Unit, Mental Health Services in the Region of Southern Denmark, Odense
  - Psychiatric Research Unit, Psychiatry, Region Sealand, Institute of Clinical Medicin, Faculty of Health Sciences, University of Copenhagen, Roskilde
- Institute of Health and Well being, University of Glasgow, Glasgow, United Kingdom

REFERENCES:
- [Derived] Stender S, Davidsen KA, Lyons-Ruth K, Harder S. Disinhibited attachment behavior among infants reared at home: Relations to maternal severe mental illness and personality disorder symptoms. Personal Disord. 2024 May;15(3):207-212. doi: 10.1037/per0000653. Epub 2024 Feb 8. PMID 38330355
- [Derived] Harder S, Davidsen K, MacBeth A, Lange T, Minnis H, Andersen MS, Simonsen E, Lundy JM, Nystrom-Hansen M, Trier CH, Rohder K, Gumley A. Wellbeing and resilience: mechanisms of transmission of health and risk in parents with complex mental health problems and their offspring--The WARM Study. BMC Psychiatry. 2015 Dec 9;15:310. doi: 10.1186/s12888-015-0692-6. PMID 26654720